CLINICAL TRIAL: NCT00996424
Title: The Effect of Inhaled N-Acetylcysteine Compared to Normal Saline on Sputum Rheology and Lung Function.
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Insufficient recruitment.
Sponsor: University Hospital, Ghent (Other)
Collaborators: BVSM (Unknown)
Responsible Party: Sabine Van Daele, MD, PhD, University Hospital Ghent
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2009/464
Record Dates: First submitted 2009-10-15; First posted 2009-10-16 (Estimated); Last update posted 2011-08-15 (Estimated); Status verified 2011-08

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — Acetylcysteine; Saline Solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acetylcysteine (Experimental): Inhalation with N-Acetylcysteine
  Interventions: Drug: Acetylcysteine
- normal saline (Placebo Comparator): Inhalation with normal saline solution
  Interventions: Drug: normal saline

INTERVENTIONS:
Drug: Acetylcysteine — Inhalation with N-Acetylcysteine
  Arms: Acetylcysteine
Drug: normal saline — Inhalation with normal saline solution
  Arms: normal saline

SUMMARY:
Inhalation treatment with mucolytics is one of the cornerstones of CF treatment for respiratory problems.

The efficacy of inhalation treatment with recombinant DNAse and hypertonic saline is well established. The North American CF foundation reported that there is insufficient evidence for or against the chronic use of inhaled N-Acetylcysteine (NAC) to improve lung function and reduce exacerbations .

In vitro tests proved the positive effect of NAC on sputum rheology . Evidence based research however on the in vivo effect of NAC on visco-elasticity and lung function is rare. There are only three randomized controlled clinical trials on nebulised NAC, none of them showing a statistically significant or clinically relevant beneficial effect. Nevertheless at least in Europe for many years inhalation treatment with NAC is advised. Because of the disgusting sulphur odour, many patients are reluctant to use this inhalation medication.

We intend to start an open placebo controlled in vivo cross-over study to evaluate the effect of Acetyl cysteine compared to normal saline on the sputum visco-elasticity and on the short term effect on lung function.

Sputum producing CF-patients, able to perform lung function tests will be enrolled.

Sputum viscoelasticity will be measured by a controlled-stress rheometer (AR 1000-N; TA-Instruments, Ghent, Belgium) at 20° C, using a cone-plate geometry 8.

Lung function measurement (FVC, FEV1, FEF 25-75) will be done in a Masterlab body plethysmograph (Jaeger®) Sputum samples will be collected before lung function test on a regular control visit. Three ml of NAC or 4 ml of normal saline will be inhaled, afterwards a second sputum sample will be collected and a control lung function test will be performed. Visco-elasticity measurements will be done on sputum samples before and after inhalation of NAC or normal saline. Patients will continue to inhale N-acetylcysteine or normal saline two times per day for one month. After one month a control lung function and a third sputum sample will be collected, visco-elasticity and lung function will be measured and compared to the initial values in both groups and between groups. After a wash-out period of normal saline inhalations during 2 weeks in both groups, patients in the initial control group will be asked to switch to inhalation of 3 ml of NAC two times per day and the former NAC group will continue to inhale two times 4 ml of normal saline during four weeks. After one month the same measurements of visco-elasticity and lung function tests will be done.

ELIGIBILITY:
Inclusion Criteria:

* Patients who can perform lung function tests and who can produce sputum (> 5 years of age)
* (Fe)males between 6-64 years

Exclusion Criteria:

* Patients on the waiting lists for lung transplant.
* Pregnancy or breast feeding
* Patients can not take part in another 'inhalation'trial for Cystic Fibrosis

Ages: 6 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 19 (Actual)
Dates: Start 2010-01; Primary Completion 2010-09 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Changes in visco-elasticity and lung function. | after one dose of N-acetylcystein compared to normal saline
Changes in visco-elasticity and lung function. | after one month of two doses per day of N-acetylcysteine compared to normal saline.

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Van Daele, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: website of the University Hospital Ghent — http://www.uzgent.be